CLINICAL TRIAL: NCT01502345
Title: Phase 1 Study to Evaluate the Safety, Tolerability, and Immunogenicity of Hantaan and Puumala Virus DNA Vaccines, pWRG/HTN-M(x) and pWRG/PUU-M(s2), for Prevention of Hemorrhagic Fever With Renal Syndrome Administered to Healthy Adult Volunteers Using the TDS-IM Electroporation Delivery Device
Brief Title: Study to Evaluate the Safety, Tolerability, and Immunogenicity of Hantaan and Puumala Virus DNA Vaccines
Acronym: HTNV/PUUV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency); United States Army Medical Materiel Development Activity (U.S. Federal Agency); Ichor Medical Systems Incorporated (Industry); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A-17088; WRAIR 1854 (Other: WRAIR IRB); S-11-12 (Other: Sponsor)
Record Dates: First submitted 2011-12-23; First posted 2011-12-30 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Hemorrhagic Fever With Renal Syndrome
Keywords: HFRS
MeSH Terms: conditions — Hemorrhagic Fever with Renal Syndrome | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- PUUV DNA Vaccine (Experimental): This group will receive Puumala Virus DNA Vaccine only
  Interventions: Biological: Vaccine/device combination for prevention of HFRS
- HTNV + PUUV (Experimental): This group will receive a 1:1 mixture of HTNV and PUUV DNA Vaccines
  Interventions: Biological: Vaccine/device combination for prevention of HFRS
- HTNV DNA Vaccine (Experimental): This group will receive Hantaan Virus DNA Vaccine only
  Interventions: Biological: Vaccine/device combination for prevention of HFRS

INTERVENTIONS:
Biological: Vaccine/device combination for prevention of HFRS — PUUV DNA Vaccine, 2.0mg/ml TDS-IM injection HTNV DNA Vaccine, 2.0 mg/ml TDS-IM injection HTNV + PUUV Vaccine mixture, 1.0mg/mL + 1.0mg/ml TDS-IM injection
  Other Names: Ichor Tri-Grid Delivery System; Hantavirus

SUMMARY:
The purpose of this study is:

• To assess safety and tolerability of the HTNV and PUUV DNA vaccines, pWRG/HTN-M(x) and pWRG/PUUV-M(s2), administered intramuscularly using a TDS-IM electroporation device

Secondary:

• To evaluate clinical immunogenicity of the HTNV and PUUV DNA vaccines, pWRG/HTN-M(x) and pWRG/PUUV-M(s2), including an assessment of the acute procedure tolerability when administered with the TDS-IM electroporation.

DETAILED DESCRIPTION:
The study will enroll 3 randomized groups of 9 subjects each, along with 3 alternates, for a total of 30 subjects. The study will include one group of subjects injected with the HTNV DNA vaccine, one group injected with the PUUV DNA vaccine, and one group injected with both HTNV and PUUV DNA vaccines (mixed), administered with the Ichor TDS-IM device. Subjects will receive one dose of vaccine on Days 0, 28, and 56 and will be followed until Day 240. Subjects will complete post-injection memory aids for 14 days after each injection.

Subjects will be evaluated for safety and immune response throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or non-pregnant, non-lactating female, ages 18-49 (inclusive) at time of screening
* Have demonstrated adequate comprehension of the protocol, by achieving a score of at least 80% correct on a short multiple-choice quiz

  * Individuals who fail to achieve a passing score on the initial quiz will be given the opportunity to retest after a review of protocol information
  * Individuals who fail the comprehension assessment for the second time will not be enrolled
* Have provided written informed consent before screening
* Free of clinically significant health problems, as determined by pertinent medical history and clinical examination before entry into the study
* Available and able to participate for all study visits and procedures
* If sexually active, known to be at least 1 year post-menopausal, or willing to use an effective method of contraception (e.g., birth control pill, diaphragm, cervical cap, intrauterine device, condom, or anatomical sterility [in self or partner]) from the date of screening until at least 6 months after the last vaccination
* Negative hantavirus IgG antibody test result at screening (ELISA)

Exclusion Criteria:

* History or serologic evidence of prior infection with either HTNV or PUUV virus, or prior participation in a HTNV or PUUV virus vaccine trial
* History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions
* Any serologic evidence of hepatitis B or C infection
* Ongoing participation in another clinical trial
* Receipt or planned receipt of any vaccination, experimental or otherwise, within the period 30 days prior to initial injection through 60 days after the Day 70 follow-up (approximately a 6 month period in total)
* Individuals in whom a skinfold measurement of the cutaneous and subcutaneous tissue for all eligible injection sites (deltoid region) exceeds 40 mm
* Individuals in whom the ability to observe possible local reactions at the eligible injection sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art
* Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, hepatic or renal functional abnormality as determined by the investigator based on medical history, physical examination, EKG, and/or laboratory screening test
* Pregnant or lactating female, or female who intends to become pregnant during the study period
* Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within 6 months of study entry

  * For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day
  * Inhaled and topical steroids are allowed
* Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child
* Syncopal episode within 12 months of screening
* Suspected or known current alcohol abuse as defined by the American Psychiatric Association in DSM IV (Diagnostic and Statistical Manual of Mental Disorders-4th edition)
* Chronic or active illicit and/or intravenous drug use
* Unwilling to allow storage and use of blood for future hantavirus-related research
* Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline for solicited adverse events after each vaccination | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14
  • The nature, frequency, and severity of local and systemic AEs or SAEs associated with TDS-IM-EP-based administration of HTNV and PUUV vaccines
Change from baseline for Unsolicited adverse events after each vaccination | Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
  • The nature, frequency, and severity of local and systemic AEs or SAEs associated with TDS-IM-EP-based administration of HTNV and PUUV vaccines

SECONDARY OUTCOMES:
Change in neutralizing antibody levels from baseline to post vaccination | Day 0, 28, 56, 84, 140, 180 and 240
  The endpoint used to measure immunogenicity of the HTNV and PUUV DNA vaccines is the production of neutralizing antibody titers to HTNV and PUUV (PRNT50 ≥ 1:20). Initial immunogenicity results will be analyzed on the basis of intention-to-treat, in which the outcomes of all subjects who had at least one dose of vaccine will be analyzed with the group to which they were originally assigned, regardless of whether they completed the study. Subsequently, all subjects who completed the 8-month study and have serologic data will be included in the analysis of immunogenicity.

CONTACTS AND LOCATIONS:
Overall Officials: James E Moon, MD, Principal Investigator — WRAIR, Clinical Trials Center
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States